CLINICAL TRIAL: NCT03107091
Title: Safety and Efficacy of Low-dose Terlipressin Delivered by Continuous Intravenous Infusion in Patients With Cirrhosis and Ascites Refractory to, or Intolerant of, Diuretic Therapy, Requiring Large Volume Paracentesis
Brief Title: Continuous Infusion Terlipressin for Patients With Cirrhosis and Refractory Ascites
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioVie Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIT-001
Record Dates: First submitted 2016-11-20; First posted 2017-04-11 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2019-04

CONDITIONS: Cirrhosis; Ascites Hepatic
Keywords: Terlipressin; Terlipressin acetate
MeSH Terms: conditions — Fibrosis | interventions — Terlipressin

STUDY DESIGN:
Intervention Model Description: Open label prospective study in a cohort of 6 patients
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Terlipressin acetate continuous infusion (Experimental): Continuous infusion of terlipressin starting at 2 mg/day over 7 days in-house and if tolerated continue treatment in the ambulatory setting for 21 days
  Interventions: Drug: Terlipressin acetate continuous infusion

INTERVENTIONS:
Drug: Terlipressin acetate continuous infusion — Low-dose continuous infusion of Terlipressin administered via ambulatory pump over 28 days
  Other Names: Terlipressin

SUMMARY:
Low-dose continuous infusion of terlipressin will be administered to six cirrhotic patients with refractory ascites.

DETAILED DESCRIPTION:
Terlipressin continuous infusion will be adminstered via an ambulatory pump initially for 7 days in a clinical pharmacology unit. Serial blood draws for pharmacokinetic analysis will be performed to determine steady state concentration of both terlipressin and 8-lysine-vasopressin during infusion. After establishing safety and tolerance of infusion for 7 days, patients will be transitioned to an outpatient setting where they will be treated with terlipressin continuous infusion for an additional 21 days, monitored daily by home care nurses.

A total of 6 patients will be treated. Monitoring will include successful management of ascites, with reduction in paracentesis procedures and decreased ascites fluid volume, further supported by improvement in renal function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis and refractory ascites who required 3 or more large volume (4 liters and more) paracenteses in the previous 60 days

Exclusion Criteria:

* Ascites with causes other than cirrhosis such as nephrogenic ascites or malignant ascites due to peritoneal carcinomatosis
* Total bilirubin > 5 mg/dL
* Blood clotting International normalized ratio (INR) > 2.5
* Serum creatinine > 2.0 mg/dL
* Current or recent (within 3 months of consent) renal dialysis
* Hepatic encephalopathy grade 3 or 4
* Superimposed acute liver failure/injury due to factors other than alcoholic hepatitis, including acute viral hepatitis, drugs, medications (e.g., acetaminophen), or other toxins (e.g., mushroom [Amanita] poisoning)
* Current or recent treatment (within 7 days) with octreotide, midodrine, vasopressin, dopamine or other vasopressors
* Respiratory failure requiring positive airway pressure devices or intubation
* SIRS/sepsis episode in the previous 28 days from consent
* Episode of spontaneous bacterial peritonitis or gastrointestinal hemorrhage within 28 days of consent
* Ongoing documented or suspected infection
* Severe cardiovascular disease that are contraindication to terlipressin therapy such as advanced arteriosclerosis, arrhythmia, coronary insufficiency or uncontrolled hypertension
* Findings suggestive of organic renal disease (severe proteinuria/hematuria, or abnormal renal ultrasound suggestive of obstructive or other renal pathology)
* Severe comorbidity that in the opinion of the Investigator would affect short-term prognosis and/or disallow safe participation in the trial (such as for example, severe anemia or pancytopenia, advanced neoplasia, hepatocellular carcinoma [confirmed with serum alpha1-fetoprotein testing], severe chronic obstructive pulmonary disease or asthma)
* Alcoholics who have not been abstinent for the past 6 months
* Transjugular intrahepatic portosystemic shunt or other surgical shunt
* For female patients: Confirmed pregnancy
* Known allergy or hypersensitivity to terlipressin
* Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yeramian, MD, Study Director — BioVie Inc.
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single site
Period: Overall Study
Arm/Group | Terlipressin Acetate Continuous Infusion
Started | 6
Completed | 5
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Terlipressin Acetate Continuous Infusion
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 61 [36 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
MELD score [Mean (Full Range); unit: score on a scale] — The Model for End-Stage Liver Disease (MELD) is a scoring system for assessing the severity of chronic liver disease and uses the subject's values for total bilirubin, serum creatinine, and the international normalized ratio (INR) for prothrombin time to predict survival. MELD is calculated according to the following formula:
  MELD = 3.78×ln[serum bilirubin (mg/dL)] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43
  The possible scores range from 6 to 40. The higher the MELD score the more severe the disease state.
  score on a scale | 15 [9 to 22]
Serum creatinine [Mean (Full Range); unit: mg/dL] | 1.30 [0.9 to 2.0]
Child-Pugh score [Mean (Full Range); unit: score on a scale] — The Pugh-Child score is determined by scoring five clinical measures of liver disease. A score of 1, 2, or 3 is given to each measure, with 3 being the most severe. The five clinical measures are: total bilirubin, serum albumin, INR, ascites and hepatic encephalopathy. The total score determines severity of disease with Class A being least severe (5-6), Class B more severe (7-9) and Class C most severe (10-15).
  score on a scale | 9 [7 to 11]

OUTCOME MEASURES:

1. Primary Outcome: Clinical Safety of Terlipressin Infusion in Cirrhotic Patients With Refractory Ascites
Description: Rate of treatment emergent adverse events assessed by physical examination and laboratory safety
Time Frame: 28 day treatment period and 28 day post-treatment
Population: Enrolled
Measure: Count of Participants; unit: Participants
Groups:
- Terlipressin Acetate Continuous Infusion: Continuous infusion of terlipressin
Arm/Group | Terlipressin Acetate Continuous Infusion
Number analyzed (Participants) | 6
Participants
  TEAE | 6
  Serious AE | 4
  Related TEAE | 3
  Serious related TEAE | 0
  TEAE leading to drug withdrawal | 3
  Grade 3 TEAE | 4
  Fatal TEAE | 0

2. Primary Outcome: Steady State Plasma Levels of Terlipressin and 8-lysine Vasopressin During Terlipressin Continuous Infusion at 2 mg/Day in Cirrhotic Patients With Refractory Ascites
Description: Serial sampling for determination of Terlipressin concentration and metabolite 8-lysine vasopressin in plasma at steady state (Css)
Time Frame: 7 day treatment
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Terlipressin Acetate Continuous Infusion
Number analyzed (Participants) | 6
ng/mL
  Terlipressin | 2.48 [1.67 to 3.23]
  8-lysine vasopressin | 0.089 [0.07 to 0.138]

3. Secondary Outcome: Change in Requirement of Large Volume Paracentesis With Continuous Infusion of Terlipressin
Description: Comparison of pre-treatment and post-treatment incidence of therapeutic paracentesis and change in volume of ascites removed
Time Frame: 28 day post-treatment
Measure: Mean (Full Range); unit: percent change
Arm/Group | Terlipressin Acetate Continuous Infusion
Number analyzed (Participants) | 6
percent change
  Percent change in volume ascites removed during 28d treatment period versus 28d pre-treatment period | -66.5 [-100.0 to -35.0]
  Percent change in LVP interval during treatment versus before treatment | 128 [0 to 414]

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | Terlipressin Acetate Continuous Infusion
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Terlipressin Acetate Continuous Infusion (N=6)
Hepatic encephalopathy (Hepatobiliary disorders) | 2 (2) — Hepatic encephalopathy
Bacteremia (Infections and infestations) | 1 (1) — Bacteremia
Ruptured umbilical hernia (Gastrointestinal disorders) | 1 (1) — Umbilical hernia
Partial bowel obstruction (Gastrointestinal disorders) | 1 (1) — Intestinal obstruction
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Terlipressin Acetate Continuous Infusion (N=6)
tachycardia (Cardiac disorders) | 1 (1) — tachycardia
diarrhea (Gastrointestinal disorders) | 1 (1) — diarrhea
Energy increased (General disorders) | 1 (1) — Increased energy
decreased appetitie (Metabolism and nutrition disorders) | 1 (1) — Decrease in appetite
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) — Hyponatremia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT03107091/Prot_SAP_000.pdf